CLINICAL TRIAL: NCT05851872
Title: A Randomized Trial of Fasting Versus Non-fasting on Outcomes and Satisfaction Prior to Cardiac Catheterization
Brief Title: Fasting Versus Non-fasting on Outcomes and Satisfaction Prior to Cardiac Catheterization
Acronym: CALORI (NPO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20025962
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (Active Comparator): Participant will be asked to fast at least 6 hours prior to the procedure
  Interventions: Procedure: Coronary angiogram; Procedure: Right heart catheterization
- Non-Fasting group (Experimental): Participants will be allowed to eat and drink up to 1 hour prior to the procedure.
  Interventions: Procedure: Coronary angiogram; Procedure: Right heart catheterization

INTERVENTIONS:
Procedure: Coronary angiogram — Being done per standard of care
Procedure: Right heart catheterization — Being done per standard of care

SUMMARY:
Moderate sedation is used in the catheterization laboratory relieve the anxiety and discomfort associated with access and other aspects of the procedure. Whether being in a fasting state (nothing per os, NPO) at the time of the procedure is beneficial or harmful is not well known, but patients are typically required to be fasting at the time of elective procedures, guidance derived from procedures that require general anesthesia. Whereas the typical thinking was that fasting prior to procedures would minimize the risk of aspiration in the event of intubation, or nausea and other symptoms generally, several studies have shown that prolonged fasting prior to procedures is associated with increased nausea, vomiting, aspiration and procedure recovery time.

We aim to evaluate patient satisfaction, nausea and immediate outcomes of patients who are not kept NPO prior to cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Requiring a cardiac catheterization as per standard of care
* Elective procedure with planned moderate sedation

Exclusion Criteria:

* BMI >45
* All emergent procedures
* All mechanical circulatory support-assisted procedures
* Other high risk procedures (as identified by the operator)
* Pregnant women
* Hemodynamically unstable patients
* Active GI illness, including nausea at the time of screening
* Taking chronic pain medications at home or on current brief course of narcotics
* Dementia
* Encephalopathy
* Patients scheduled for deep sedation
* Severe GERD (if the patient requires more than one medication for adequate control of GERD symptoms or has required medical intervention within the past year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Pre-procedure wellness score (hunger, tiredness, anxiety, nausea) | Baseline (Prior to procedure)
  We get a wellness score prior to the procedure (right before the patient is taken into the lab) and is on a 0-5 scale with 0 being very happy and 5 being very unhappy.
Intra- and post-procedural vomiting, aspiration, and intubation checklist | Within 24 hours after the procedure
  We review the chart and ask the participant if they had any vomiting. We also review the chart to see if there are any reports/concern of aspiration and follow up on any chest X-rays that were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Gertz, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be considered upon each individual request.
Supporting Information: Study Protocol
Time Frame: Data sharing will be considered upon each individual request.
Access Criteria: Data sharing will be considered upon each individual request.